CLINICAL TRIAL: NCT03014362
Title: Utility of Repetitive Transcranial Magnetic Stimulation (TMS) in Promoting Rapid Psychiatric Stabilization in Acutely Suicidal Military Service Members
Brief Title: TMS for Suicidal Crisis in Active Duty SMs
Acronym: TMS4SI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eisenhower Army Medical Center (U.S. Federal Agency)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Augusta University (Other); The Geneva Foundation (Other)
Responsible Party: Principal Investigator, Christopher Hines, Chief, DDEAMC Outpatient Behavioral Health, Eisenhower Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1604023
Record Dates: First submitted 2016-11-30; First posted 2017-01-09 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Suicide; Suicidal Ideation; Suicidal Impulses; Suicidal Intention; Suicidal and Self-Injurious Behavior; Suicidal Depression
MeSH Terms: conditions — Suicide; Suicidal Ideation; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TMS active (Active Comparator): Neuronetics NeuroStar XPLOR magnetic stimulator - Active;
  Localization: Left prefrontal dorsolateral neocortex. Dose Delivery: Figure-8 solid core coil at 120% motor threshold, 10 Hz, 4 second train duration, 10 second interval for 30 minutes.
  Treatment Dose: ~4k/session, 12-15k/day, 36-45k total pulses. Sessions: 9 in total; 3/day for 3 consecutive days over and above SOC (Standard of Care).
  Interventions: Device: Neuronetics NeuroStar XPLOR magnetic stimulator - Active
- TMS sham (Sham Comparator): Neuronetics NeuroStar XPLOR magnetic stimulator - Sham;
  Localization: Left prefrontal dorsolateral neocortex. Sham Delivery: Figure-8 solid core coil rendered inert via blocking insert. Dose: Zero pulses. Sessions: 9 in total; 3/day for 3 consecutive days over and above SOC.
  Interventions: Device: Neuronetics NeuroStar XPLOR magnetic stimulator - Sham

INTERVENTIONS:
Device: Neuronetics NeuroStar XPLOR magnetic stimulator - Active — Localization: Left prefrontal dorsolateral neocortex. Dose Delivery: Figure-8 solid core coil at 120% motor threshold, 10 Hz, 4 second train duration, 10 second interval for 30 minutes.
  Treatment Dose: ~4k/session, 12-15k/day, 36-45k total pulses. Sessions: 9 in total; 3/day for 3 consecutive days over and above SOC.
  Arms: TMS active
Device: Neuronetics NeuroStar XPLOR magnetic stimulator - Sham — Localization: Left prefrontal dorsolateral neocortex. Sham Delivery: Figure-8 solid core coil rendered inert via blocking insert. Dose: Zero pulses. Sessions: 9 in total; 3/day for 3 consecutive days over and above SOC.
  Arms: TMS sham

SUMMARY:
The purpose of this study is to determine if the use of Transcranial Magnetic Stimulation (TMS) provides rapid reduction and sustained attenuation of suicidal crisis. TMS is a treatment for suicidal crisis that is quicker, less invasive, better tolerated, and with fewer side effects than current treatments such as Electroconvulsive Therapy (ECT) and medication therapies. There will be 6 months of follow-up, in order to establish the ongoing and lasting therapeutic effect of TMS.

DETAILED DESCRIPTION:
The programmatic-level objective of the study is to address the goals of the Army STARRS Program and the Suicide Prevention for America's Veterans Act through implementation of an effective acute treatment for patients psychiatrically admitted in suicidal crisis as well as other patients at high-risk for suicide. This is achieved by application of TMS, which provides a treatment for suicidal crisis that is quicker, less invasive, better tolerated, and with fewer side effects and less incapacitation than current treatments such as ECT and pharmacologic therapies. A recent study led by the senior consultant of this proposal demonstrated tolerance and efficacy for a new, high-dose regimen of TMS in a VA population with an average age of 47. The objective of the proposed study is to extend the application of TMS to a younger population of Active Duty Service Members (SM) in order to demonstrate efficacy for returning veterans of the Middle East wars, in particular, as well as the civilian young adult population. TMS dosage in the proposed study is recalibrated to commercially-standard levels in order to provide consistency with devices currently in clinical operation. In addition, follow-up in the proposed study continues for 6 months in order to establish persistence and durability of the therapeutic effect of TMS.

ELIGIBILITY:
Inclusion Criteria:

* All Active Duty SMs (regardless of sex, ethnicity, sexual or religious orientation) who are admitted to Eisenhower Army Medical Center (EAMC) Inpatient Psychiatric Service (IPS) with active suicidality or elevated risk for suicide regardless of most psychiatric diagnostic co-morbidity (see exclusion criteria). This includes in-patient admissions for suicidality and outpatient SMs with a Columbia-Suicide Severity Rating Scale (C-SSRS) score ≥3.
* Age 18 to 60
* Able to speak and read English.

Exclusion Criteria:

* Combative with staff.
* Comatose/catatonia.
* Incapacity owing to active mania or psychosis.
* Epilepsy, multiple sclerosis, or cerebrovascular accident.
* Non-removable metal in the head (Shrapnel; plates, aneurysm coils/clips; metal tattoos etc.)
* Implantable devices (pacemakers, stimulators, etc.)
* Schizophrenic or borderline personality.
* Positive screen for pregnancy.
* Already receiving TMS as a treatment for depression.
* Non-English reading and speaking subjects

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Hines, MD, Principal Investigator — Eisenhower Army Medical Center
Locations (1):
- Eisenhower Army Medical Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hines CE, Mooney S, Watson NL, Looney SW, Wilkie DJ. Repetitive Transcranial Magnetic Stimulation Promotes Rapid Psychiatric Stabilization in Acutely Suicidal Military Service Members. J ECT. 2022 Jun 1;38(2):103-109. doi: 10.1097/YCT.0000000000000810. PMID 35613009

RESULTS

PARTICIPANT FLOW:
Groups:
- TMSactive: TMSactive
- TMSsham: TMSsham
Period: Overall Study
Arm/Group | TMSactive | TMSsham
Started | 59 | 61
Completed (completed) | 41 | 51
Not Completed | 18 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMSactive | TMSsham | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 61 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (6.9) | 26.5 (6.4) | 27.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 44 | 42 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  demographic: black | 8 | 13 | 21
  demographic: white | 35 | 39 | 74
  demographic: hispanic | 10 | 5 | 15
  demographic: other | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 59 | 61 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change in Suicidal Ideation (Acute)
Description: The Beck Scale for Suicidal Ideation (SSI-T) is a 19-item clinician administered scale measuring current suicide ideation (SSI-C), suicide ideation at its worst point in the patient's life (SSI-W), and degree of hopelessness. The scale has been well validated. SSI-T scores range from 0-38, with higher scores indicating greater suicide risk.
Time Frame: Change over the active treatment course ie. the 3 days of active treatment
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- TMS Active: Group receiving active treatment
- TMSsham: group receiving sham treatment
Arm/Group | TMS Active | TMSsham
Number analyzed (Participants) | 59 | 61
score on a scale | 0.12 (0.06) | 0.12 (0.06)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- TMS Sham: group receiving sham treatment
Arm/Group | TMS Active | TMS Sham
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/61
Serious Adverse Events (participants affected / at risk) | 2/59 | 2/61
Other Adverse Events (participants affected / at risk) | 18/59 | 7/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Active (N=59) | TMS Sham (N=61)
suicidal ideation (Psychiatric disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Active (N=59) | TMS Sham (N=61)
pain (Psychiatric disorders) | 18 (18) | 7 (7) — Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03014362/Prot_007.pdf
  • Statistical Analysis Plan (2020-08-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT03014362/SAP_005.pdf